CLINICAL TRIAL: NCT04687462
Title: Comparison of 1-mm Thickness Variance Polyethylene Insert Total Knee Arthroplasty System and 2-mm Thickness Variance Polyethylene Insert Total Knee Arthroplasty System in the Same Patients
Brief Title: Comparison of Polyethylene Insert Variances of Different Total Knee Arthroplasty System in the Same Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC20DISI0965
Record Dates: First submitted 2020-12-10; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Total Knee Replacement Arthroplasty

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-centered, randomized controlled clinical trial. Patients undergoing bilateral total knee replacement arthroplasty(TKRA) for both knee osteoarthritis will receive written consent from the patient through informed consent before the surgery. Among the patients undergoing total arthroplasty for both knee joints, only patients who have agreed with written consent will receive the surgery. In one patient who has been decided to be erolled for the stedy, we will set one knee joint as the experimental group, and the other knee joint as the control group. The experimental group will undergo TKRA using Exult total knee system and the control group will get TKRA using Lospa total knee system.
Who Masked: Participant
Masking Description: The researcher performing the surgery can know which instruments are used for each knee joint according to the random number table assignment result, but the subjects undergoing surgery will be conducted as a single blinded study where it is not possible to know which instruments are used for each side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): TKRA operation undergoing 1-mm thickness variance polyethylene insert total knee arthroplasty system (Exult, Corentec)
  Interventions: Device: 1-mm thickness variance polyethylene insert total knee arthroplasty system (Exult, Corentec)
- Control (Active Comparator): TKRA operation undergoing 2-mm thickness variance polyethylene insert total knee arthroplasty system (Lospa, Corentec)
  Interventions: Device: 1-mm thickness variance polyethylene insert total knee arthroplasty system (Exult, Corentec)

INTERVENTIONS:
Device: 1-mm thickness variance polyethylene insert total knee arthroplasty system (Exult, Corentec) — TKRA operation undergoing 1-mm thickness variance polyethylene insert total knee arthroplasty system (Exult, Corentec)

SUMMARY:
Total knee arthroplasty(TKA) is a successful orthopedic surgery with excellent clinical outcome and survival. However, there are concerns about patient satisfaction in previous reports, and dissatisfaction rate of 15-30% is reported in clinical outcomes(PROMs) of some studies. Therefore, for improving the patient's outcome and satisfaction after total knee arthroplasty, it is necessary to change the design of the conventional total knee arthroplsaty implant. The knee is a joint structure with several dynamic functions, and not only the skeletal structure but also the soft tissue balance plays an important role in the function of the knee joint. New implants are being developed to overcome the limitations of conventional TKA implant, including the Exult total knee system (Exult; Corentec). Exult implant has 1mm thickness variance of polyethylene insert, which is different from the conventional total knee systems. This new total knee system has been shown in experimental studies to produce nearly normal knee movement.

The clinical results of this more specific variance of polyethyelen insert thickness total knee implant system are insufficient, and there is also a lack of comparative studies with conventional total knee arthroplasty implant. The purpose of this study is to compare outcomes between 1-mm thickness variance polyethylene insert total knee arthroplasty system(Exult, total knee system, Corentec) and conventional 2-mm thickness variance polyethylene insert total knee arthroplasty system(Lospa total knee system, Corentec) in the same patients. This study is a randomized controlled study in patients undergoing both knee total knee arthroplasty in a day. Radiologic parameter, patients preference and clinical results was investigated in both knee of same patients who received TKA during minimum 2 year follow up.

DETAILED DESCRIPTION:
This study is a prospective, single-centered, randomized controlled clinical trial. Patients undergoing bilateral total knee replacement arthroplasty(TKRA) for both knee osteoarthritis will receive written consent from the patient through informed consent before the surgery. Among the patients undergoing total arthroplasty for both knee joints, only patients who have agreed with written consent will receive the surgery. In one patient who has been decided to be erolled for the stedy, we will set one knee joint as the experimental group, and the other knee joint as the control group. The experimental group will undergo TKRA using Exult total knee system and the control group will get TKRA using Lospa total knee system. The researcher performing the surgery can know which instruments are used for each knee joint according to the random number table assignment result, but the subjects undergoing surgery will be conducted as a single blinded study where it is not possible to know which instruments are used for each side.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis patients for both total knee arthroplasty
* having medicare insurance

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Crystal-induced arthritis
* Septic arthritis
* Neuropsychiatric patients
* Previous knee operation history
* Patients with preoperative severe limitation of motion (Flexion ontracture ≥ 20, range of motion ≤ 90)
* Patients with preoperative severe defomity of knee alignment (Varus or valgus angle ≥ 15)
* Severe obese patients (BMI ≥ 40)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Arthritis Index(WOMAC) pain scale | Preoperative & postoperative 3, 6, 12, 24 months
  Changes of post-operative WOMAC score from pre-operative WOMAC scores at post-operative 3, 6, 12, 24 months WOMAC score ranges (0 ~ 96 in total score)

SECONDARY OUTCOMES:
Knee Society Score | Preoperative & postoperative 3, 6, 12, 24 months
  Changes of post-operative Knee Society Score from pre-operative Knee Society Score scores at post-operative 3, 6, 12, 24 months KSS score ranges (0 ~ 150 in total score)
Knee range of motion | Preoperative & postoperative 3, 6, 12, 24 months
  Changes of post-operative knee ROM from pre-operative knee ROM at post-operative 3, 6, 12, 24 months (normal knee full range motion is 0 degree to 135 degrees in flexion)

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Principal Investigator — the Catholic Univerisity of Korea Seoul St Mary's hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR